CLINICAL TRIAL: NCT05244447
Title: Imperial Valley Regional Occupational Program (IVROP) ReadyforLIFE Healthy Marriage and Responsible Fatherhood Program Evaluation
Brief Title: IVROP ReadyforLIFE Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Imperial Valley Regional Occupational Program (IVROP) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/38
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Youth

STUDY DESIGN:
Intervention Model Description: Arms Primary services: Participants receive 12 hours of Relationships Smarts Plus, 3 hours of Mind Matters and 1 hour of Money Habitudes workshops over the course of 10 weeks. Participants also receive life coaching and ongoing job readiness support.
  Assigned Interventions Primary services: Participants receive 12 hours of Relationships Smarts Plus, 3 hours of Mind Matters and 1 hour of Money Habitudes workshops over the course of 10 weeks. Participants also receive life coaching and ongoing job readiness support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Services (Experimental): Primary services: Participants receive 12 hours of Relationships Smarts Plus, 3 hours of Mind Matters and 1 hour of Money Habitudes workshops over the course of 6 weeks. Participants also receive life coaching and on-going job readiness support.
  Interventions: Other: Primary Services

INTERVENTIONS:
Other: Primary Services — Primary services: Participants receive 12 hours of Relationships Smarts Plus, 3 hours of Mind Matters and 1 hour of Money Habitudes workshops over the course of 6 weeks. Participants also receive life coaching and ongoing job readiness support.

SUMMARY:
The purpose of the Imperial Valley Regional Occupational Program (IVROP) ReadyforLIFE program evaluation is to determine whether primary (i.e., behaviors) and secondary (i.e., attitudes) outcomes improve for youth participants after completing the ReadyforLIFE program. Understanding the ways in which the IVROP ReadyforLIFE program supports healthy partner relationships and economic stability is important for those providing services to at-risk youth populations.

DETAILED DESCRIPTION:
After being informed about the study and giving consent, participants will enroll in a program that collects data at enrollment, at the end of the program, and 12 months following program enrollment. The length of the program ranges from four weeks up to one year, depending on the setting and the number of optional workshops students opt to receive. Research questions in this study are framed by a descriptive evaluation design to assess whether outcomes improve for at-risk youth who participate in the IVROP ReadyforLIFE program. Primary and secondary outcomes are assessed before and one year after participants complete core curricula - Relationships Smart Plus, Mind Matters, and Money Habitudes (pre to follow-up). Primary outcome measures will indicate whether behavior improved for healthy partner relationships and financial stability. Secondary outcome measures will indicate whether improvements were made in the attitudes and expectations that facilitate and reflect behavior for healthy partner relationships and financial stability.

ELIGIBILITY:
Inclusion Criteria:

* At-risk youth (foster/justice involved, immigrant household, undocumented, LGBTQ)
* High school age
* Residing in the Imperial Valley, CA

Exclusion Criteria:

* Individuals who are 18 and above and out of high school
* Individuals who reside outside of Imperial Valley, CA

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1054 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- Imperial Valley Regional Occupational Program Community Foundation (IVROPCF), El Centro, California, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Services
Started | 1054
Completed | 1054
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Services
Number analyzed (Participants) | 1054
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1006
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.2 [13 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 526
  Male | 528
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 976
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 29
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 35
  Black or African American | 4
  White | 405
  More than one race | 476
  Unknown or Not Reported | 93

OUTCOME MEASURES:

1. Primary Outcome: Healthy Partner Relationship Behavior Measurement #1
Description: Will participants report significantly healthier relationship behaviors one year after enrolling into the IVROP ReadyforLIFE program?
  Items measured include:
  5 items: levels of reported skill with key relationship behaviors (categories, 4-point scale); measured on the Healthy Relationship Behavior Scale #1 as:
  1 = I am extremely good at this 2 = I am good at this 3 = I am bad at this 4 = I am extremely bad at this Lower scores indicate a higher perceived skill in healthy relationship behaviors, so the lower the rating, the better the score.
  The 5 items are measured as a construct. All items are added together and divided by 5 to create the construct score. The lower the score, the better the outcome.
  maximum score of 4.0, minimum score of 1.0.
Time Frame: Change from baseline in behavior in relationship behavior (interaction with romantic partner at 12 months from enrollment
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 516
score on scale
  Mean at baseline | 2.93 (.4847)
  Mean at follow-up | 2.97 (.4834)

2. Primary Outcome: Healthy Partner Relationship Behavior Measurement #2
Description: 1B) Will participants report significantly healthier relationship behaviors one year after enrolling into the IVROP ReadyforLIFE program?
  Items measured include:
  6 items: frequency of engaging in key relationship behaviors (categories, 5-point scale); measured on the Healthy Relationship Behavior Scale #2 as:
  1 = None of the time 2 = Some of the time 3 = Half of the time 4 = Most of the time 5 = All of the time
  Higher scores indicate a higher perceived frequency of engaging in unhealthy relationship behaviors, so the higher the rating, the worse the score.
  Reverse scoring will have the higher score always equal to showing improvement.
  The 6 items are measured as a construct. All items are added together and divided by 6 to create the construct score. The lower the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: change from baseline in behavior to 12-months after program completion
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 160
score on scale
  Mean at baseline | 4.17 (.562)
  Mean at follow-up | 4.14 (.584)

3. Primary Outcome: Money Management Scale (Financial Behavior Measurement #1)
Description: Will participants report significantly healthier financial behavior one year after enrolling into the IVROP ReadyforLIFE program?
  Items measured include:
  4 items: frequency of engaging in healthy money management behaviors (categories, 5-point scale); measured on the Money Management Scale #1 as:
  1 = Never 2 = Rarely 3 = Sometimes 4 = Often 5 = Always Higher scores indicate a greater frequency of engaging in healthy money management behaviors, so the higher the rating, the better the score.
  The 4 items are measured as a construct. All items are added together and divided by 4 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: change from baseline in behavior to 12-months after program completion
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 744
score on scale
  Mean at baseline | 3.45 (.861)
  Mean at follow-up | 3.54 (.830)

4. Secondary Outcome: Healthy Partner Relationship Attitudes Measurement #1
Description: Will participants report significantly healthier partner relationship attitudes one year after enrolling into the IVROP ReadyforLIFE program?
  Items measured include:
  9 items: levels of agreement with relationship beliefs (categories, 4-point); measured on the Healthy Relationship Attitudes #1 Scale as:
  1 = Strongly Agree 2 = Agree 3 = Disagree 4 = Strongly Disagree Higher scores indicate a higher disagreement with unhealthy relationship attitudes, so the higher the rating, the better the score.
  The 9 items are measured as a construct. All items are added together and divided by 9 to create the construct score. The higher the score, the better the outcome.
  maximum score of 4.0, minimum score of 1.0.
Time Frame: change from baseline in behavior to 12-months after program completion
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 823
score on scale
  Mean at baseline | 2.36 (.376)
  Mean at follow-up | 2.40 (.403)

5. Secondary Outcome: Healthy Partner Relationship Attitudes Measurement #2
Description: Will participants report significantly healthier partner relationship attitudes one year after enrolling into the IVROP ReadyforLIFE program?
  Items measured include:
  3 items: future-oriented self-reported beliefs in key relationship events likely to occur (categories, 5-point scale); measured on the Healthy Partner Relationship Attitudes Measurement #2 as:
  1 = Almost no chance 2 = Some chance but probably not 3 = A 50-50 chance 4 = A good chance 5 = Almost certain Higher scores indicate a greater perceived likelihood of key relationship events to occur in the future. Two items will be reverse coded so that for all items, a higher rating will indicate a better score.
  The 3 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0.
Time Frame: change from baseline in behavior to 12-months after program completion
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 810
score on scale
  Mean at baseline | 3.45 (.646)
  Mean at follow-up | 3.45 (.632)

6. Secondary Outcome: Financial Attitudes Measurement #1
Description: Do participants report significantly healthier financial attitudes one year after enrolling into the IVROP ReadyforLIFE program?
  Items measured include:
  7 items: levels of agreement with key financial attitudes (categories, 5-point scale); measured on the Financial Attitudes Scale as:
  1 = Strongly Disagree 2 = Disagree 3 = Neither Agree nor Disagree 4 = Agree 5 = Strongly Agree Higher scores indicate a higher positive attitude towards healthy financial management, so the higher the rating, the better the score.
  The 7 items are measured as a construct. All items are added together and divided by 7 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0.
Time Frame: change from baseline in behavior to 12-months after program completion
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 709
score on scale
  Mean at baseline | 3.71 (.516)
  Mean at follow-up | 3.69 (.541)

ADVERSE EVENTS:
Time Frame: 1 year through study completion
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Primary Services
All-Cause Mortality (participants affected / at risk) | 0/1054
Serious Adverse Events (participants affected / at risk) | 0/1054
Other Adverse Events (participants affected / at risk) | 0/1054

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT05244447/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT05244447/SAP_001.pdf